CLINICAL TRIAL: NCT02294643
Title: A Multicenter Randomized Trial Evaluating the Efficacy of Sarpogrelate on Ischemic Heart Disease After Drug-eluting Stent Implantation in Patients With Diabetes Mellitus or Renal Impairment
Brief Title: Study Design of 'Influence of Sarpogrelate in Patients With Renal Impairment or Diabetes Mellitus' Study
Acronym: SERENADE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Yuhan Corporation (Industry)
Responsible Party: Principal Investigator, Dong-Ju Choi, Chief of Cardiovascular Center in Seoul National University Bundang Hospital, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SERENADE trial
Record Dates: First submitted 2014-11-10; First posted 2014-11-19 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Coronary Artery Disease; Diabetes Mellitus; Renal Insufficiency, Chronic
Keywords: sarpogrelate
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus; Renal Insufficiency, Chronic | interventions — sarpogrelate; Aspirin; Clopidogrel; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- aspirin, clopidogrel & sarpogrelate (Active Comparator): the triple anti-platelet treatment group will receive aspirin 100mg, clopidogrel 75mg and sarpogrelate (Anplag®, Yuhan Corporation, Seoul, South Korea) 100mg twice daily
  Interventions: Drug: Sarpogrelate; Drug: Aspirin; Drug: Clopidogrel
- aspirin, clopidogrel & placebo (Placebo Comparator): the dual anti-platelet group will receive aspirin 100mg and clopidogrel 75mg daily plus placebo twice daily
  Interventions: Drug: Aspirin; Drug: Clopidogrel; Drug: Placebo (for Sarpogrelate)

INTERVENTIONS:
Drug: Sarpogrelate
  Other Names: Anplag
  Arms: aspirin, clopidogrel & sarpogrelate
Drug: Aspirin
  Other Names: Astrix; Aspirin protect
Drug: Clopidogrel
  Other Names: Plavix
Drug: Placebo (for Sarpogrelate)
  Other Names: sugar pill manufactured to mimic sarpogrelate tablet
  Arms: aspirin, clopidogrel & placebo

SUMMARY:
The purpose of the SERENADE trial is to evaluate the safety and efficacy of sarpogrelate in patients with CKD or DM after DES implantation.

DETAILED DESCRIPTION:
The rates of stent failure after percutaneous intervention (PCI) have declined after introduction of the drug eluting stent (DES). However, chronic kidney disease (CKD) or diabetes mellitus (DM) still remains a strong clinical predictor of poor prognosis with DES. Sarpogrelate, a selective 5-HT2a receptor antagonist, has antiproliferative effects as shown by its reduction of neointimal hyperplasia and smooth muscle cell proliferation as well as a potent antiplatelet agent inhibiting of 5-HT-induced platelet aggregation. However, the efficacy and safety data for sarpogrelate in patients with CKD or DM are limited. We aimed to test whether sarpogrelate has beneficial effects in patients with CDK or DM treated with DES.

The SERENADE trial is a multicenter, off-label, prospective, placebo-controlled randomized study to test the superiority of triple anti-platelet therapy (TAT; aspirin, clopidogrel and sarpogrelate) to the conventional dual antiplatelet therapy (DAT; aspirin and clopidogrel) in preventing late lumen loss 9 months after the index procedure in patients with CKD or DM. A total of 220 patients exhibiting coronary artery disease (CAD) with DM or CKD will be randomized to TAT or DAT (1:1 ratio) after DES implantation. Primary endpoint is late lumen loss at 9 months assessed by quantitative coronary angiography (QCA). Secondary efficacy endpoints are composites of major adverse cardiovascular events (MACE) including cardiac death, nonfatal myocardial infarction (MI), and target lesion revascularization. Secondary safety endpoints are major bleeding event and hepatic or renal impairments.

The SERENADE trial will give insight whether adjunctive therapy with sarpogrelate is helpful for patients with high risk profiles such as CKD or DM after DES implantation.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic CAD (including acute coronary syndrome) or positive stress test and a native coronary lesion (>50% diameter stenosis by visual estimation on coronary angiogram and reference diameter > 2.5 mm)
* AND CKD or DM patients

Exclusion Criteria:

* if they had contraindication to aspirin, clopidogrel or sarpogrelate.

Min Age: 18 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2009-04; Primary Completion 2012-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
late lumen loss measured by quantitative coronary angiography | 9 months

SECONDARY OUTCOMES:
all cause deaths | 12 months
cardiac death | 12 months
nonfatal myocardial infraction | 12 months
target lesion revascularization | 12 months
major bleeding using the TMI bleeding classification | 12 months
hepatic impairments as measured by ncreased serum glutamyl oxaloacetic transaminase level or glutamyl pyruvic transaminase level increased more than threefold of the upper normal range | 12 months
  increased serum glutamyl oxaloacetic transaminase level or glutamyl pyruvic transaminase level increased more than threefold of the upper normal range
renal impairments as measured by increased microalbuminuria or decreased creatinine clearance | 12 months
  increased microalbuminuria or decreased creatinine clearance

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, South Korea

REFERENCES:
- [Derived] Natale P, Palmer SC, Saglimbene VM, Ruospo M, Razavian M, Craig JC, Jardine MJ, Webster AC, Strippoli GF. Antiplatelet agents for chronic kidney disease. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD008834. doi: 10.1002/14651858.CD008834.pub4. PMID 35224730
- [Derived] Lee SA, Suh JW, Park JJ, Yoon CH, Cho YS, Youn TJ, Chae IH, Kim HS, Kim SH, Choi DJ. Study design of the influence of SErotonin inhibition on patients with RENAl impairment or diabetes undergoing drug-eluting stent implantation (SERENADE) study: A multicenter, open-label, prospective, randomized study. Contemp Clin Trials. 2015 Jul;43:20-4. doi: 10.1016/j.cct.2015.04.005. Epub 2015 Apr 16. PMID 25891091